CLINICAL TRIAL: NCT05189041
Title: Determination of the Aneurysm Vulnerability Index by Stimulation and Medical Imaging
Acronym: ANEUVISM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9364
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Aneurysm
Keywords: aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruptured Cerebral Aneurysm (Other): Quantify the aneurysmal pulsation in functional MRI on the patient with Ruptured Cerebral Aneurysm
  Interventions: Other: Aneurysmal pulsation in functional MRI
- Non Ruptured Cerebral Aneurysm (Other): Quantify the aneurysmal pulsation in functional MRI on the patient with Non Ruptured Cerebral Aneurysm
  Interventions: Other: Aneurysmal pulsation in functional MRI

INTERVENTIONS:
Other: Aneurysmal pulsation in functional MRI — Quantify the aneurysmal pulsation in functional MRI on the patient with Ruptured Cerebral Aneurysm

SUMMARY:
Stroke is the leading cause of disability in France with 130,000 cases per year, 20% of strokes being hemorrhagic, with a majority of intracranial aneurysm rupture (80%). Each year, 6000 meningeal hemorrhages (MHA) caused by cerebral aneurysm rupture are reported in France: 40% of patients die within the first month and 30% are left with severe and permanent disability. Intracranial aneurysms are present in 2 to 6% of the population and only about 0.5% of them will rupture. Given the human and economic costs associated with this disease, systematic medical screening for intracranial aneurysms could be useful. However, the operative risk of endovascular treatment remains non-zero (around 1%) and could be proposed only to a selected population of aneurysms at risk of rupture. The absence of diagnostic criteria for aneurysmal vulnerability does not allow for the moment to consider screening for this disease, which continues to strike without warning a young and active population.

Nevertheless, access to brain imaging allows the detection of an increasing number of intracranial aneurysms. The question of preventive treatment then arises and is still a difficult point discussed by neurosurgeons / neurointerventionists based on general epidemiological data difficult to apply to an individual.

ELIGIBILITY:
Inclusion Criteria:

* Age limits to > 18 years
* Collection of the informed consent (patient or legal representant)
* Affiliation or recipient with the mode of social security

  - Groupe anévrysme rompu
* Patient porteur d'un anévrysme rompu

  - Groupe anévrysme non rompu
* Patient porteur d'un anévrysme non rompu

Exclusion Criteria:

* Subject presenting contraindications in MRI (Ferromagnetic foreign bodies, pace-maker …)
* Claustrophobia
* Women pregnant or Breast-feeding
* Patient participating in an other study
* Patient have participated in a study in the 3 months before the inclusion
* In period of exclusion relative to another protocol
* Person with majority age protected by the law (supervision or trusteeship).
* Patient not reading the french language
* Patient or representant for whom it impossible to give accurate informations

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Quantify the aneurysmal pulsation in functional MRI | 1 day
  Quantify the aneurysmal pulsation in functional MRI on the patient with Ruptured Cerebral Aneurysm or Non ruptured Aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT COSTALAT, Study Director — University Hospital, Montpellier
Locations (1):
- COSTALAT, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided